CLINICAL TRIAL: NCT01870518
Title: Neurocognitive Effects of Bilateral Subthalamic Nucleus Versus Globus Pallidus Interna Deep Brain Stimulation in Parkinson's Disease Patients With Mild Cognitive Impairment
Brief Title: Neurocognitive Effects of Bilateral STN Versus GPi DBS in Parkinson's Disease Patients With MCI
Acronym: DBS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13BN006
Record Dates: First submitted 2013-05-01; First posted 2013-06-06 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Parkinson's Disease; Mild Cognitive Impairment; Dementia
Keywords: Parkinson's disease; Dementia
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parkinson's patients with MCI (Active Comparator): Procedure: deep brain stimulation surgery
  Interventions: Device: Bilateral GPi DBS; Device: Bilateral STN DBS
- Parkinson's patients without MCI (Active Comparator): Procedure: deep brain stimulation surgery
  Interventions: Device: Bilateral GPi DBS; Device: Bilateral STN DBS

INTERVENTIONS:
Device: Bilateral GPi DBS
Device: Bilateral STN DBS

SUMMARY:
Purpose: This is a prospective single-center, randomized, patient and evaluator-blind clinical trial to compare the neurocognitive outcomes of globus pallidus interna (GPi) versus subthalamic nucleus (STN) deep brain stimulation (DBS) in Parkinson's disease (PD) patients with mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) of the globus pallidus interna (GPi) or subthalamic nucleus (STN) has been accepted as the surgical treatment of choice for patients with advanced Parkinson's Disease (PD), demonstrating improvements in motor function that exceed those achieved by medical management alone. Unfortunately, a paucity of data exist comparing non-motor outcomes between DBS of the available targets. Specifically, a high prevalence of concurrent cognitive dysfunction or early dementia exists in PD patients, and it is unclear whether DBS target selection may have differential effects with regards to cognitive outcomes in PD patients with early evidence of mild cognitive impairment Previous studies indicate that stimulation of either the GPi or STN is associated with decrements in patients' verbal fluency, visuospatial memory, as well as overall cognitive decline, but those patients were randomized without consideration for baseline neurocognitive performance and it is unclear whether these effects are due to treatment or rather the natural history of these patients.

In addition to the clinical arm of this trial, another secondary goal is to evaluate several biomarkers obtained from blood and cerebrospinal in order to determine their utility if any as prognosticators of patient cognitive and motor outcomes. Specifically, we will be evaluating levels of amyloid 1-42, total tau, phosphorylated tau 181, and brain derived neurotrophic factor in the cerebrospinal fluid as well as genotyping the apolipoprotein-E gene. These proteins and genotypes are still currently under investigation as potential biomarkers for dementia as well as neuroplasticity.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of idiopathic Parkinson's disease
* deemed an appropriate candidate for DBS surgery
* Montreal Cognitive Assessment (MoCA) score < 25
* Neuropsychological testing with the diagnosis of Mild Cognitive Impairment

Exclusion Criteria:

* no diagnosis of Parkinson's disease
* not appropriate for DBS surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Neurocognitive Function | 6 months post-operative
  By focusing on patients with MCI, our primary aim will be to detect whether STN or GPi DBS incur target specific impacts on patients' subsequent neurocognitive function.Patients will undergo neuropsychological testing pre-operatively and again at six months post-operatively. Patient's will also undergo a Montreal Cognitive Assessment at specified intervals: pre-operatively, 3weeks, 6 weeks and 6 months post-operatively.

SECONDARY OUTCOMES:
Functional motor improvements | 6 month post-operative
  The secondary aim will be measure functional motor outcomes in our patients.Patient's will undergo Unified Parkinson's Disease Rating Scale (UPDRS 3 and 4) motor testing pre-operatively in the off medication and on medication states. Patients will be re-tested 6 months post-operatively in the following states: on device / off medication, off device / off medication, on device / on medication.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco A Ponce, MD, Principal Investigator — Barrow Neurological Institute / St. Joseph's Hospital & Medical Center
Locations (1):
- Barrow Neurological Institute / St. Joseph's Hospital & Medical Center, Phoenix, Arizona, United States

REFERENCES:
- [Background] Weaver FM, Follett KA, Stern M, Luo P, Harris CL, Hur K, Marks WJ Jr, Rothlind J, Sagher O, Moy C, Pahwa R, Burchiel K, Hogarth P, Lai EC, Duda JE, Holloway K, Samii A, Horn S, Bronstein JM, Stoner G, Starr PA, Simpson R, Baltuch G, De Salles A, Huang GD, Reda DJ; CSP 468 Study Group. Randomized trial of deep brain stimulation for Parkinson disease: thirty-six-month outcomes. Neurology. 2012 Jul 3;79(1):55-65. doi: 10.1212/WNL.0b013e31825dcdc1. Epub 2012 Jun 20. PMID 22722632
- [Background] Aarsland D, Zaccai J, Brayne C. A systematic review of prevalence studies of dementia in Parkinson's disease. Mov Disord. 2005 Oct;20(10):1255-63. doi: 10.1002/mds.20527. PMID 16041803
- [Background] Rodriguez-Oroz MC, Obeso JA, Lang AE, Houeto JL, Pollak P, Rehncrona S, Kulisevsky J, Albanese A, Volkmann J, Hariz MI, Quinn NP, Speelman JD, Guridi J, Zamarbide I, Gironell A, Molet J, Pascual-Sedano B, Pidoux B, Bonnet AM, Agid Y, Xie J, Benabid AL, Lozano AM, Saint-Cyr J, Romito L, Contarino MF, Scerrati M, Fraix V, Van Blercom N. Bilateral deep brain stimulation in Parkinson's disease: a multicentre study with 4 years follow-up. Brain. 2005 Oct;128(Pt 10):2240-9. doi: 10.1093/brain/awh571. Epub 2005 Jun 23. PMID 15975946
- [Background] Follett KA, Weaver FM, Stern M, Hur K, Harris CL, Luo P, Marks WJ Jr, Rothlind J, Sagher O, Moy C, Pahwa R, Burchiel K, Hogarth P, Lai EC, Duda JE, Holloway K, Samii A, Horn S, Bronstein JM, Stoner G, Starr PA, Simpson R, Baltuch G, De Salles A, Huang GD, Reda DJ; CSP 468 Study Group. Pallidal versus subthalamic deep-brain stimulation for Parkinson's disease. N Engl J Med. 2010 Jun 3;362(22):2077-91. doi: 10.1056/NEJMoa0907083. PMID 20519680
- [Background] Mayeux R, Saunders AM, Shea S, Mirra S, Evans D, Roses AD, Hyman BT, Crain B, Tang MX, Phelps CH. Utility of the apolipoprotein E genotype in the diagnosis of Alzheimer's disease. Alzheimer's Disease Centers Consortium on Apolipoprotein E and Alzheimer's Disease. N Engl J Med. 1998 Feb 19;338(8):506-11. doi: 10.1056/NEJM199802193380804. PMID 9468467
- [Background] Hansson O, Buchhave P, Zetterberg H, Blennow K, Minthon L, Warkentin S. Combined rCBF and CSF biomarkers predict progression from mild cognitive impairment to Alzheimer's disease. Neurobiol Aging. 2009 Feb;30(2):165-73. doi: 10.1016/j.neurobiolaging.2007.06.009. Epub 2007 Jul 23. PMID 17646035
- [Background] Park H, Poo MM. Neurotrophin regulation of neural circuit development and function. Nat Rev Neurosci. 2013 Jan;14(1):7-23. doi: 10.1038/nrn3379. PMID 23254191